CLINICAL TRIAL: NCT05248269
Title: Safety and Efficacy of Stereo-Electroencephalography Guided Thermocoagulation in Drug Resistant Focal Epilepsy
Brief Title: Thermocoagulation in Drug Resistant Focal Epilepsy
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: State Budgetary Healthcare Institution, National Medical Surgical Center N.A. N.I. Pirogov, Ministry of Health of Russia (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NMSC-01-22
Record Dates: First submitted 2022-02-04; First posted 2022-02-21 (Actual); Last update posted 2024-07-23 (Actual); Status verified 2024-07

CONDITIONS: Epilepsy; Seizures, Focal; Epilepsy Intractable; Epilepsies, Partial
MeSH Terms: conditions — Epilepsy; Seizures; Drug Resistant Epilepsy; Epilepsies, Partial

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Thermocoagulation of epileptogenic zone (Experimental)
  Interventions: Procedure: Radiofrequency thermocoagulation

INTERVENTIONS:
Procedure: Radiofrequency thermocoagulation — The 2 pertinent contacts connect to Radiofrequency thermocoagulation lesion-generator equipment (Cosman G4 with Ad-tech electrodes), expressly modified for use with SEEG electrodes. The following parameters will be adopted: current power 3 W within 180 seconds and current intensity (usually approximately 25 mA) variable according to impedance.

SUMMARY:
Therapeutic thermocoagulation will be carried out in patients with drug-resistant focal epilepsy in cases where an epileptogenic zone is found and proven according to stereo-electroencephalography (SEEG) data.

DETAILED DESCRIPTION:
Open-label, pilot, non-comparative, interventional cohort study. Each patient will be examined at least 8 times (8 visits will pass): Visit 0 - screening (within 14 days before Visit 1), Visit 1 (visit includes the procedure for the destruction of the epileptogenic focus), Visits 2 and 3 (after 1 and 2 days after Visit 1) - a repeated procedure for the destruction of the epileptogenic focus with an incomplete effect of the first procedure (not mandatory, carried out by the decision of the principal investigator), Visits 4-7 (7, 14, 30, 180 days after the procedure for the destruction of the epileptogenic focus).

Patients will be divided into 4 cohorts of 4 patients. Enrollment in the study of the next cohort of patients will be based on the safety analysis of the previous cohort 1 day after the manipulation.

After assessing the position of the electrodes based on the conjugation of brain MRI data before and after SEEG implantation and seizure recording, the ictal zone is determined. Thus, the localization of pathological activity is determined on the basis of neuroimaging data, as well as in accordance with the activity under certain contacts of the SEEG electrodes.

After explaining the treatment options to the patient and relatives, informed voluntary consent is taken for the implementation of this procedure.

Using a radio frequency generator Cosman RFG-G4, destruction is carried out at the necessary electrode contacts with a power of 3W, exposure time of 180 sec. In case of pain occurrence, the procedure is immediately terminated. After the procedure, the patient continues SEEG monitoring for 3 days.

If additional epileptogenic zones are identified, if necessary, a repeated thermocoagulation is performed (on the 2nd and 3rd days of the study). If there is no need for a second thermocoagulation, then Visits 2 and 3 are not performed. Next, the patient undergoes removal of the electrodes, a control MRI study is performed. Follow-up includes follow-up for 6 months. Visits 4-6 involve phone interviews with patients. During the conversation, the researcher should clarify complaints, general well-being, the presence and frequency of epileptic seizures over the period of time that has passed since the previous visit.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of symptomatic drug-resistant epilepsy according to anamnesis, results of video EEG monitoring with registration of epileptic seizures.
2. The epileptogenic zone verified using invasive electrodes.
3. The patient has read the information sheet and signed the informed consent form.

Non-inclusion Criteria:

1. Persons with mental disorders.
2. Women during pregnancy, childbirth.
3. Women during breastfeeding.
4. Reception of anticoagulants.
5. Location of the epileptogenic focus within functionally significant areas, large vessels of the brain.
6. Primary generalized forms of epilepsy.

Exclusion Criteria:

1. Absence of a registered seizure on stereo-EEG.
2. Absence of a focal pattern during invasive stereo-EEG monitoring.

Dropout Criteria:

1. Refusal of the patient from observation
2. The occurrence of contraindications that may prevent participation in diagnostic and treatment activities.
3. Unwillingness or inability of the patient to comply with the requirements of the protocol, including the presence of any condition (physical, mental or social) that may affect his ability to comply with the requirements of the study
4. Identification of conditions during the study that meet the exclusion criteria for non-inclusion of patients.
5. Lack of effect from thermocoagulation within a month after manipulation or worsening of the condition associated with an increase in the number/severity of epileptic seizures.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 75 (Actual)
Dates: Start 2022-02-07 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Severe adverse reactions and events rate | Up to 6 months after procedure
  Severe adverse reactions and events will be monitored and registered during procedure of thermocoagulation and up to 6 months after procedure
Seizure freedom or reduction after procedure | Up to 6 months after procedure
  The incidence of seizures will be assessed and registered daily by patient in the diary for self-inspection. Records in the diary will be inspected by investigators during follow-up visits.

SECONDARY OUTCOMES:
Three-level European quality of life five-dimensional questionnaire | Up to 6 months after procedure
  There are five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 3 levels: no problems, some problems, and extreme problems. Patients choice results into a 1-digit number that expresses the level selected for that dimension. The digits for the five dimensions can be combined into a 5-digit number that describe the health status.
Pittsburgh Sleep Quality Index (PSQI) Questionnaire | Up to 6 months after procedure
  The Pittsburgh Sleep Quality Index (PSQI) is a questionnaire that assesses sleep quality over a 1 month time frame. It consists of 19 individual elements, making up 7 components that give one overall rating. Each item is weighted on a scale from 0 to 3. The overall PSQI score is then calculated by adding the scores of the seven components to give an overall score of 0 to 21, where lower scores mean healthier sleep quality.
Change of epileptiform activity on electroencephalography (EEG) study | Days 1, 7, 180
  EEG will be registered and reduction of epileptiform activity will be assessed (Beta, Theta, spikes, sharp waves).
Beck Depression Inventory | Up to 6 months after procedure
  This is a 21-question test that helps determine the psychological state of a person.
  The score for each category is calculated as follows: each item on the scale is scored from 0 to 3 according to the increasing severity of the symptom. The total score ranges from 0 to 63 and decreases as the condition improves.
  The questionnaire is handed out to the patient and filled out by him independently.
  The results are evaluated depending on the number of points scored:
  0-13 - variations considered normal 14-19 - mild depression 20-28 - moderate depression 29-63 - severe depression

CONTACTS AND LOCATIONS:
Overall Officials: Andrey A Zuev, MD, PhD, Principal Investigator — Pirogov National Medical and Surgical Center
Locations (1):
- Pirogov National Medical and Surgical Center, Moscow, Russia

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: CSR
Time Frame: 2 months after completion of the study
Access Criteria: upon the request